CLINICAL TRIAL: NCT06651021
Title: A Phase I, Open-label Study to Assess the Pharmacokinetics, Safety and Tolerability Following Administration of a Single Dose of Balcinrenone/Dapagliflozin in Healthy Chinese Participants
Brief Title: A Phase I PK Study of Balcinrenone/Dapagliflozin in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6402C00014
Record Dates: First submitted 2024-09-25; First posted 2024-10-21 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteer
Keywords: Chinese Healthy Volunteer; Phase 1; Pharmacokinetics; Safety; Tolerability; balcinrenone/dapagliflozin
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- balcinrenone/dapagliflozin (Experimental): To evaluate the PK of balcinrenone /dapagliflozin given as a single dose to healthy Chinese participants
  Interventions: Drug: balcinrenone/dapagliflozin

INTERVENTIONS:
Drug: balcinrenone/dapagliflozin — Each participant will receive a single dose of balcinrenone/dapagliflozin 40 mg/10 mg capsule on Day 1 under fasted condition.
  Each participant will be involved in the study for up to 35 days.

SUMMARY:
This study is intended to evaluate the PK, safety, and tolerability of balcinrenone/dapagliflozin given as a single dose capsule to healthy Chinese participants.

DETAILED DESCRIPTION:
This is a Phase I, open-label, single-arm, single dose PK study in healthy Chinese participants to be conducted at a single study centre in mainland China. In this study, approximately 10 participants (both females and males) will be assigned to the IMP. Each participant will receive a single dose of a capsule with balcinrenone/dapagliflozin 40 mg/10 mg on Day 1 under fasted condition. The study will comprise of the following:

* A screening period
* A treatment period
* A follow-up visit At the discretion of the investigator, the participant may remain in the study center until the completion of the follow-up visit

ELIGIBILITY:
Inclusion Criteria:

Age

1. Participant aged 18 to 50 years.

   Type of Participant and Disease Characteristics
2. Chinese participants who are healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.

   Weight
3. Body weight within 50.0-100.0 kg and BMI within the range 19.0-28.0 kg/m2 (inclusive) at screening.

Exclusion Criteria:

Medical Conditions

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the administration of IMP.
4. Any clinically significant abnormal findings in vital signs, as judged by the investigator.
5. Any clinically important abnormalities in clinical chemistry, haematology or urinalysis results as judged by the investigator.
6. Any positive result on screening for serum HBsAg or anti-hepatitis B core antibody, hepatitis C antibody, and HIV antibody.
7. Positive screen for drugs of abuse, alcohol or cotinine at screening or on admission to the study centre.
8. Suspected or confirmed COVID-19 infection within the last 4 weeks prior to screening or admission. Or hospitalisation for COVID-19 within the last 12 weeks prior to screening or admission.
9. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
10. Current smokers or those who have smoked or used nicotine products within the 3 months prior to screening.
11. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to balcinrenone or dapagliflozin.

    Prior/Concomitant Therapy
12. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), hormone replacement therapy, herbal remedies, megadose vitamins and minerals within 14 days or 5 half-lives (whichever is longer) before the start of IMP, unless, in the opinion of the investigator, the medication will not interfere with the study.

    Prior/Concurrent another Clinical Study Experience
13. Has received investigational product within 3 months (or 5 half-lives, whichever is longer) of administration of study intervention in this study.

    Other Exclusions
14. Involvement in the planning and/or conduct of this study.
15. Judgment by the investigator that the participant should not participate in this study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
16. Previous enrolment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
AUCinf of AUCinf of balcinrenone/dapagliflozin | Day 1 to post dose 48 hours
  To evaluate the PK of balcinrenone /dapagliflozin given as a single dose to healthy Chinese participants
AUClast of balcinrenone /dapagliflozin | Day 1 to post dose 48 hours
  To evaluate the PK of balcinrenone /dapagliflozin given as a single dose to healthy Chinese participants
Cmax of balcinrenone /dapagliflozin | Day 1 to post dose 48 hours
  To evaluate the PK of balcinrenone /dapagliflozin given as a single dose to healthy Chinese participants
C24h of balcinrenone /dapagliflozin | Day 1 to post dose 48 hours
  To evaluate the PK of balcinrenone /dapagliflozin given as a single dose to healthy Chinese participants
tmax of balcinrenone /dapagliflozin | Day 1 to post dose 48 hours
  To evaluate the PK of balcinrenone /dapagliflozin given as a single dose to healthy Chinese participants
t½λz of balcinrenone /dapagliflozin | Day 1 to post dose 48 hours
  To evaluate the PK of balcinrenone /dapagliflozin given as a single dose to healthy Chinese participants
λz of balcinrenone /dapagliflozin | Day 1 to post dose 48 hours
  To evaluate the PK of balcinrenone /dapagliflozin given as a single dose to healthy Chinese participants
CL/F of balcinrenone /dapagliflozin | Day 1 to post dose 48 hours
  To evaluate the PK of balcinrenone /dapagliflozin given as a single dose to healthy Chinese participants
MRTinf of balcinrenone /dapagliflozin | Day 1 to post dose 48 hours
  To evaluate the PK of balcinrenone /dapagliflozin given as a single dose to healthy Chinese participants
Vz/F of balcinrenone /dapagliflozin | Day 1 to post dose 48 hours
  To evaluate the PK of balcinrenone /dapagliflozin given as a single dose to healthy Chinese participants

OTHER OUTCOMES:
Incidence of AEs and SAEs | From ICF throughout the treatment period and including the follow-up period (7 days post-dose）
  To assess the safety and tolerability of balcinrenone/dapagliflozin given as a single dose to healthy Chinese participants
Incidence of abnormal Supine blood pressure | From ICF throughout the treatment period and including the follow-up period (7 days post-dose）
  To assess the safety and tolerability of balcinrenone/dapagliflozin given as a single dose to healthy Chinese participants
Incidence of abnormal Supine Pulse | From ICF throughout the treatment period and including the follow-up period (7 days post-dose）
  To assess the safety and tolerability of balcinrenone/dapagliflozin given as a single dose to healthy Chinese participants
Height in centimeter | From ICF throughout the treatment period and including the follow-up period (7 days post-dose）
  This is related to Body Mass Index, To assess the safety and tolerability of balcinrenone/dapagliflozin given as a single dose to healthy Chinese participants
Weight in Kilograms | From ICF throughout the treatment period and including the follow-up period (7 days post-dose）
  This is related to Body Mass Index, To assess the safety and tolerability of balcinrenone/dapagliflozin given as a single dose to healthy Chinese participants
Incidence of abnormal clinical chemistry assessments：Glucose, HbA1c, Creatinine, , ALP, ALP, ALT, AST, total bilirubin, Potassium, Chloride, Bicarbonate, Calcium (total), magnesium, Phosphorous, Sodium, CK, eGFR, FSH, hCG | From ICF throughout the treatment period and including the follow-up period (7 days post-dose）
  To assess the safety and tolerability of balcinrenone/dapagliflozin given as a single dose to healthy Chinese participants
Incidence of abnormal urinalysis: Glucose, Haemoglobin, Protein/Albumin, hCG | From ICF throughout the treatment period and including the follow-up period (7 days post-dose）
  To assess the safety and tolerability of balcinrenone/dapagliflozin given as a single dose to healthy Chinese participants
Incidence of abnormal haematology assessments: Haematocrit, Hb, Platelet count, RBC, WBC | From ICF throughout the treatment period and including the follow-up period (7 days post-dose）
  To assess the safety and tolerability of balcinrenone/dapagliflozin given as a single dose to healthy Chinese participants
Incidence of abnormal of Electrocardiogram parameter: ECG mean heart rate | From ICF throughout the treatment period and including the follow-up period (7 days post-dose）
  To assess the safety and tolerability of balcinrenone/dapagliflozin given as a single dose to healthy Chinese participants
Incidence of abnormal of Electrocardiogram parameter: ECG Heart rhythm | From ICF throughout the treatment period and including the follow-up period (7 days post-dose）
  To assess the safety and tolerability of balcinrenone/dapagliflozin given as a single dose to healthy Chinese participants
Incidence of abnormal of Electrocardiogram parameter: ECG QRS duration, QT interval, QTc interval Fridericia | From ICF throughout the treatment period and including the follow-up period (7 days post-dose）
  To assess the safety and tolerability of balcinrenone/dapagliflozin given as a single dose to healthy Chinese participants
Incidence of abnormal physical examination: assessments of general appearance, respiratory, CV, abdomen, neurological systems, the skin, lymph nodes | From ICF throughout the treatment period and including the follow-up period (7 days post-dose）
  To assess the safety and tolerability of balcinrenone/dapagliflozin given as a single dose to healthy Chinese participants
Incidence of abnormal physical examination: assessment of the presence and extent of peripheral (ankle/leg) oedema | From ICF throughout the treatment period and including the follow-up period (7 days post-dose）
  To assess the safety and tolerability of balcinrenone/dapagliflozin given as a single dose to healthy Chinese participants

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Chengdu, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
  Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home